CLINICAL TRIAL: NCT03721341
Title: A Randomized Phase III Trial of Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of 4-10 Oligometastatic Tumors (SABR-COMET 10)
Brief Title: Stereotactic Ablative Radiotherapy for Comprehensive Treatment of 4-10 Oligometastatic Tumors
Acronym: SABR-COMET 10
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: David Palma (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); British Columbia Cancer - Centre for the North (Unknown); Beaston West of Scotland Cancer Centre (Unknown); London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABR-COMET 10
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Drug Therapy; Immunotherapy; Hormones; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard arm (Active Comparator): Standard of care treatment: palliative radiotherapy, chemotherapy, immunotherapy, hormones, or observation, is at the discretion of the treating oncologist.
  Interventions: Radiation: Palliative Radiation; Drug: Chemotherapy; Drug: Immunotherapy; Drug: Hormones; Other: Observation
- Stereotactic Arm (Experimental): Stereotactic ablative radiotherapy, plus standard of care treatment: chemotherapy, immunotherapy, hormones, or observation given at the discretion of the treating oncologist.
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy; Drug: Hormones; Other: Observation; Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Palliative Radiation — Investigators should follow the principles of palliative radiotherapy as per the individual institution in order to alleviate symptoms or prevent complications. If radiotherapy is indicated, recommended doses are 8 Gy in 1 fraction, 20 Gy in 5 fractions, and 30 Gy in 10 fractions.
  Other Names: Palliative Radiotherapy
  Arms: Standard arm
Drug: Chemotherapy — Chemotherapy may be given as indicated.
Drug: Immunotherapy — Immunotherapy may be given as indicated.
Drug: Hormones — Hormones may be given as indicated.
Other: Observation — Observation only is acceptable if this is the standard practice.
Radiation: Stereotactic Ablative Radiotherapy — Total dose of radiation and number of fractions will depend on the site of disease. Doses are 20 Gy in 1 fraction, 30 Gy in 3 fractions (every 2 days), or 35 Gy in 5 fractions (daily).
  Arms: Stereotactic Arm

SUMMARY:
In patients with a limited oligometastatic burden (cancer has spread but is not yet considered metastatic), emerging evidence suggests that treatment of all sites of disease with ablative therapies can improve patient outcomes, including overall- and progression-free survival. The application of Stereotactic Ablative Radiotherapy (SABR) for patients with 4-10 metastatic deposits appears promising, yet it is unclear if all patients with greater than 3 oligometastatic lesions benefit from ablative therapies in terms of improved Overall Survival (OS), Progression Free Survival (PFS), or quality of life. The purpose of this study is to assess the impact of SABR, compared to standard of care treatment, on overall survival, oncologic outcomes, and quality of life in patients with a controlled primary tumor and 4-10 metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* Karnofsky performance score greater than 60
* Life expectancy greater than 6 months
* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* Controlled primary tumor defined as: at least 3 months since original tumor treated definitively, with no progression at primary site
* Total number of metastases 4-10
* All sites of disease can be safely treated based on a pre-plan

Exclusion Criteria:

* Serious medical comorbidities precluding radiotherapy. These include interstitial lung disease in patients requiring thoracic radiation, Crohn's disease in patients where the GI tract will receive radiotherapy, and connective tissue disorders such as lupus or scleroderma.
* For patients with liver metastases, moderate/severe liver dysfunction (Child Pugh B or C)
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated with radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed below. All such cases must be discussed with one of the study PIs.
* Malignant pleural effusion
* Inability to treat all sites of disease
* Any single metastasis greater than 5 cm in size.
* Any brain metastasis greater than 3 cm in size or a total volume of brain metastases greater than 30 cc.
* Metastasis in the brainstem
* Clinical or radiologic evidence of spinal cord compression
* Dominant brain metastasis requiring surgical decompression
* Metastatic disease that invades any of the following: GI tract (including esophagus, stomach, small or large bowel), mesenteric lymph nodes, or skin
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival at Study Completion | At approximately end of year 6 (study completion)
  Time from randomization to death from any cause.

SECONDARY OUTCOMES:
Progression-free Survival | At approximately year 3, and end of year 6 (study completion)
  Time from randomization to disease progression at any site or death.
Time from randomization to development of new metastatic lesions | At approximately end of year 6 (study completion)
  New metastatic lesions will be detected using computed tomography, magnetic resonance imaging, and/or bone scans.
Quality of Life as measured by the Functional Assessment of Cancer Therapy- General (FACT-G) questionnaire | At approximately end of year 6 (study completion)
Quality of Life as measured by the EuroQOL Group EQ-5D-5L questionnaire | At approximately end of year 6 (study completion)
Toxicity as measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | End of years 1, 2, 3, 4, 5, and 6 (study completion)
Overall Survival at midpoint of Study | At approximately year 3 (midpoint)

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, Principal Investigator — London Health Sciences Centre, Lawson Health Research Institute; Suresh Senan, MRCP, FRCR, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Robert Olson, MD, Principal Investigator — British Columbia Cancer - Centre for the North; Stephen Harrow, MB ChB, Principal Investigator — Beaston West of Scotland Cancer Centre
Locations (14):
- Alfred Health, Melbourne, Victoria, Australia
- Canada (9):
  - BC Cancer Agency, Vancouver Island Centre, Victoria, British Columbia
  - Nova Scotia Health Authortiy, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Trillium Health Partners-Credit Valley Hospital, Mississauga, Ontario
  - Niagra Health System, St. Catharines, Ontario
  - University Health Network, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal-CHUM, Montreal, Quebec
- VU University Medical Centre, Amsterdam, Netherlands
- University Hospital of Zürich, Zurich, Switzerland
- United Kingdom (2):
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mattes MD, Eubank TD, Almubarak M, Wen S, Marano GD, Jacobson GM, Ma PC. A Prospective Trial Evaluating the Safety and Systemic Response From the Concurrent Use of Radiation Therapy with Checkpoint Inhibitor Immunotherapy in Metastatic Non-Small Cell Lung Cancer. Clin Lung Cancer. 2021 Jul;22(4):268-273. doi: 10.1016/j.cllc.2021.01.012. Epub 2021 Jan 25. PMID 33608212
- [Derived] Palma DA, Olson R, Harrow S, Correa RJM, Schneiders F, Haasbeek CJA, Rodrigues GB, Lock M, Yaremko BP, Bauman GS, Ahmad B, Schellenberg D, Liu M, Gaede S, Laba J, Mulroy L, Senthi S, Louie AV, Swaminath A, Chalmers A, Warner A, Slotman BJ, de Gruijl TD, Allan A, Senan S. Stereotactic ablative radiotherapy for the comprehensive treatment of 4-10 oligometastatic tumors (SABR-COMET-10): study protocol for a randomized phase III trial. BMC Cancer. 2019 Aug 19;19(1):816. doi: 10.1186/s12885-019-5977-6. PMID 31426760